CLINICAL TRIAL: NCT00588016
Title: Concentration of Itraconazole Solution in Nasal Secretions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hirohito Kita, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-009651
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Sinusitis
Keywords: Itraconazole
MeSH Terms: conditions — Sinusitis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Itraconazole (Experimental): Topical application of Itraconazole in Sterile Water 100 mg/1000 ml, irrigating each nostril with 20 ml of solution twice daily for 7 days.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Topical application of Itraconazole in Sterile Water 100 mg/1000 ml, irrigating each nostril with 20 ml of solution twice daily for 7 days.
  Other Names: Sporanox

SUMMARY:
The primary objective of this study is to determine the concentration of itraconazole irrigation in nasal mucous specimens via collection and High-performance liquid chromatography (HPLC) assay.

Eight (8) patients with chronic rhinosinusitis (CRS) and two (2) healthy controls will be enrolled in the initial evaluation. After an initial control nasal specimen, followed by seven days of twice daily topical itraconazole irrigation, nasal specimens will be collected at varying time intervals and the concentrations measured.

The primary endpoint is development of a reliable collection and assay technique with concentration curves over time of topically administered itraconazole. A secondary endpoint is to determine if the concentrations measured achieve a mean inhibitory concentration (MIC90) to commonly cultured fungal species in the nose.

DETAILED DESCRIPTION:
This is a pilot study for the purpose of gathering concentration data on a commonly used topical antifungal solution of itraconazole. CRS patients that meet the defined inclusion criteria will begin topical itraconazole antifungal irrigations on Day 1. This will consist of Itraconazole in Sterile Water 100 mg/1000 ml, irrigating each nostril with 20 ml of solution twice daily, with a bulb syringe as directed. The patient will return on Day 7 for repeat examination and nasal secretion collection. Two patients will be randomly selected to have blood drawn at the completion of day 7 testing to determine the concentration of itraconazole in the blood.

ELIGIBILITY:
Inclusion Criteria:

General:

* Greater than or equal to eighteen years of age.
* Patient must be willing to be available and comply with all scheduled procedures as defined in the protocol.
* Patients that have been felt to be candidates for topical itraconazole therapy and would have been started on the therapy regardless of study inclusion

Medical:

* CRS defined by American Academy of Otolaryngology - Head and Neck Surgery (AAO HNS) guidelines

Controls:

* Do not meet CRS definitions. No acute sinusitis within past 4 weeks. No previous surgery for rhinosinusitis. No history of allergic rhinitis or other rhinologic disorders.

Exclusion Criteria:

General:

* Previous use of a topical antifungal nasal irrigation within the past 2 weeks or a systemic antifungal medication within the past 3 months.

Medical:

* History of cystic fibrosis, immunodeficiency, immotile cilia syndrome, clinical or radiographic suspicion for fungal mycetoma or invasive fungal sinusitis
* Pregnancy - female patients of child bearing age will undergo a pregnancy test, if positive they will be excluded
* History of liver disease
* History of congestive heart failure
* Allergy or sensitivity to itraconazole, or other azole antifungals, or any other ingredient in the preparation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Concentration of Itraconazole in nasal secretions at 7 days | 7 days after initiation of study

CONTACTS AND LOCATIONS:
Overall Officials: Hirohito Kita, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States